CLINICAL TRIAL: NCT02814565
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Multicenter Trial to Study the Efficacy and Safety of Cyclobenzaprine HCl Extended Release (CER) 15 mg in Subjects With Acute Cervical and/or Lower Back Pain Due to Muscle Spasms of Local Origin
Brief Title: Cyclobenzaprine HCl Extended Release 15 mg Versus Placebo in Treatment of Cervical and/or Lower Back Pain Due to Muscle Spasms of Local Origin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYC-RR-001; U1111-1162-4846 (Registry Identifier: WHO)
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-01

CONDITIONS: Neck Pain; Back Pain; Spasm
Keywords: Drug therapy
MeSH Terms: conditions — Neck Pain; Back Pain; Spasm | interventions — cyclobenzaprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclobenzaprine HCl 15 mg (Experimental): Cyclobenzaprine Hydrochloride (HCl) extended-release, 15 mg capsules, orally, once daily for 14 days.
  Interventions: Drug: Cyclobenzaprine HCl
- Placebo (Placebo Comparator): Cyclobenzaprine HCl extended release placebo-matching capsules, orally, once daily for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclobenzaprine HCl — Cyclobenzaprine HCl extended-release capsules
  Other Names: Myorix®; AMRIX®
  Arms: Cyclobenzaprine HCl 15 mg
Drug: Placebo — Cyclobenzaprine HCl extended release placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the effect of cyclobenzaprine hydrochloride (HCl) extended release (CER) 15 mg capsule once daily in participants with muscle spasms associated with acute painful musculoskeletal conditions.

DETAILED DESCRIPTION:
The drug being tested in this study was cyclobenzaprine hydrochloride (HCl) extended-release (CER). CER was being tested to treat participants who had muscle spasms associated with acute painful musculoskeletal conditions. This study looked at medication helpfulness, relief from muscle spasms and pain, and improvement in range of motion and daily living activities.

The study enrolled 180 participants. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups which remained undisclosed to the participant and study doctor during the study:

* CER 15 mg
* Placebo (dummy inactive pill) - this was a capsule that looks like the study drug but had no active ingredient

All participants were asked to take one capsule at the same time each day throughout the study.

This multi-center trial was conducted in the Russian Federation. The overall time to participate in this study was up to 45 days. Participants made multiple visits to the clinic, and were contacted by telephone after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is experiencing for no more than 14 days cervical or lower back pain (as assessed by the participant) due to muscle spasms (confirmed by the physician) associated with acute, painful musculoskeletal conditions.
4. Is male or female and aged 18 to 50 years, inclusive.
5. Female participants require to be either 2 years postmenopausal or surgically sterile by bilateral tubal ligation, hysterectomy, or bilateral oophorectomy, or, if premenopausal, had to be using an approved contraceptive method.
6. Female participants of child-bearing potential must have a negative urine human chorionic gonadotropin (hCG) test result for pregnancy at study entry.
7. After signing the informed consent form, the participant agrees not to make changes to dietary, exercise, or smoking habits and not to enter a weight loss program during his/her participation in the study.

Exclusion Criteria:

1. Has muscular pain secondary to acute trauma or fractures (e.g., due to osteoporosis). Such conditions could have been ruled out based on medical history, x-ray, or physical examination.
2. Has received any investigational compound within 30 days prior to Screening.
3. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
4. Has a history of drug abuse or recent (within the last 12 months) history of excessive alcohol consumption defined as >2 drinks/day (>90 ml of 80 proof alcohol or equivalent).
5. Has mild, moderate, severe liver impairment.
6. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
7. Takes any concomitant medication including over-the-counter and herbal products for muscle spasms. If a participant is taking such medications, the medications has to be discontinued before starting the study.
8. Takes or took within last 14 days medications, such as:

   1. selective serotonin reuptake inhibitors (SSRIs);
   2. serotonin norepinephrine reuptake inhibitors (SNRIs);
   3. tricyclic antidepressants (TCAs);
   4. monoamine oxidase (MAO) inhibitors;
   5. tramadol;
   6. bupropion;
   7. meperidine;
   8. verapamil;
   9. non-steroid anti-inflammatory drugs (NSAIDs);
   10. topical anti-inflammatory medications
9. Has a history or clinical manifestations of significant medical condition, such as:

   1. hyperthyroidism;
   2. acute recovery phase of myocardial infarction;
   3. arrhythmias, heart block or conduction disturbances;
   4. congestive heart failure;
   5. angle-closure glaucoma;
   6. urinary retention;
   7. increased intraocular pressure.
10. Has abnormal physical findings or a medical condition that might have placed the participant at risk or interfered with the participant's ability to participate in the study.
11. Has any known condition or disorder that might have affected absorption of the study drug.
12. Has a history of hypersensitivity or allergies to cyclobenzaprine and/or tricyclic antidepressants or any of their components.
13. Has a history of hypersensitivity to any NSAIDs including salicylate sensitivity.
14. Has a history of thrombocytopenia.
15. Has a history of gastro-intestinal bleeding, cerebrovascular bleeding or other bleeding disorders.
16. Had active or history of recurrent peptic ulcer/haemorrhage (two or more distinct episodes of proven ulceration or bleeding)
17. Has a history of severe renal impairment
18. Had a major surgery during the 6 months preceding study entry.
19. Has a language barrier or any other problems precluding good communication or cooperation.
20. Has any reason to believe that he/she would not be able to complete the evaluations needed in this study.
21. Has a known history of positive screen for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) antibody.
22. Drug abuse in anamnesis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (10):
- Russia (10):
  - Lipetsk, Lipetsk Oblast
  - Saransk, Respublika Mordoviya
  - Yekaterinburg, Sverdlovsk Oblast
  - Kazan', Tatarstan Republic
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Saint Petersburg
  - Tver'
  - Yaroslavl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in the Russian Federation from 12 October 2016 to 14 March 2017.
Pre-assignment Details: Participants with a diagnosis of acute cervical and/or lower back pain due to muscle spasms of local origin were enrolled equally in one of two treatment groups: Cyclobenzaprine HCl 15 mg or placebo.
Period: Overall Study
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo
Started | 90 | 90
Completed | 89 | 88
Not Completed | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Subject decision, caused by AE Influenza | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included participants who received at least one dose of investigation product, analyzed according to original treatment assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (9.0) | 31.5 (9.2) | 32.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 62 | 110
  Male | 42 | 28 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  European (Caucasian) | 90 | 90 | 180
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 90 | 90 | 180
Smoking Status [Count of Participants; unit: Participants]
  Never smoked | 78 | 79 | 157
  Former smoker | 1 | 3 | 4
  Current smoker | 11 | 8 | 19
Height [Mean (Standard Deviation); unit: cm] | 171.8 (8.2) | 169.1 (7.6) | 170.5 (8.0)
Weight [Mean (Standard Deviation); unit: kg] | 71.05 (14.53) | 66.22 (13.61) | 68.64 (14.25)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Subject's Rating of Medication Helpfulness Impression on Day 3 of Treatment
Description: Participants assessed the study medication helpfulness on a daily basis (in the daily diary), using the following 5-point rating scale: "How would you rate this study medication in improving your condition?" "0 = poor", "1 = fair", "2 = good", "3 = very good", "4 = excellent".
Time Frame: Day 3
Population: FAS included participants who received at least one dose of investigation product, analyzed according to original treatment assignment.
Measure: Number; unit: percentage of participants
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo
Number analyzed (Participants) | 90 | 90
percentage of participants
  Day 3, 0=poor | 20.0 | 28.9
  Day 3, 1=fair | 60.0 | 46.7
  Day 3, 2=good | 16.7 | 22.2
  Day 3, 3=very good | 3.3 | 2.2
  Day 3, 4=excellent | 0.0 | 0.0
Statistical Analysis 1: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; The 2-sample Wilcoxon rank sum test was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 0.05 level of significance; Test type: Superiority; p = 0.6179, Wilcoxon Rank Sum test

2. Secondary Outcome: Percentage of Participants With Subject's Rating of Medication Helpfulness Impression on Days 7 and 14 of Treatment
Description: as for outcome 1
Time Frame: Days 7 and 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo
Number analyzed (Participants) | 90 | 90
percentage of participants
  Day 7, 0=poor | 7.8 | 16.7
  Day 7, 1=fair | 41.1 | 34.4
  Day 7, 2=good | 35.6 | 34.4
  Day 7, 3=very good | 13.3 | 11.1
  Day 7, 4=excellent | 2.2 | 3.3
  Day 14, 0=poor | 8.9 | 14.4
  Day 14, 1=fair | 25.6 | 25.6
  Day 14, 2=good | 25.6 | 28.9
  Day 14, 3=very good | 22.2 | 20.0
  Day 14, 4=excellent | 17.8 | 11.1
Statistical Analysis 1: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; Day 7. The 2-sample Wilcoxon rank sum test was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 0.05 level of significance; Test type: Superiority; p = 0.4338, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; Day 14. The 2-sample Wilcoxon rank sum test was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 0.05 level of significance; Test type: Superiority; p = 0.1657, Wilcoxon Rank Sum Test

3. Secondary Outcome: Percentage of Participants With Physician's Clinical Global Assessment on Day 3 of Treatment
Description: The investigator assessed their clinical global impression of change compared to Baseline, based on physical examination, degree of muscle spasm (presence of muscle spasm assessment), reaction to palpation (presence of local pain assessment), limitation of range of motion, and evaluation of the patient's reported functional assessment (limitation of activities of daily living assessment). The following 5-point rating scale was used: "1 = worse", "2 = no change", "3 = slight improvement", "4 = moderate improvement", "5 = marked improvement".
Time Frame: Day 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo
Number analyzed (Participants) | 90 | 90
percentage of participants
  Day 3, 1=worse | 1.1 | 0.0
  Day 3, 2=no change | 52.2 | 68.9
  Day 3, 3=slight improvement | 35.6 | 25.6
  Day 3, 4=moderate improvement | 11.1 | 3.3
  Day 3, 5=marked improvement | 0.0 | 2.2
Statistical Analysis 1: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; The 2-sample Wilcoxon sum rank test was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 0.05 level of significance; Test type: Superiority; p = 0.0393, Wilcoxon Sum Rank Test

4. Secondary Outcome: Percentage of Participants With Physician's Clinical Global Assessment on Days 7 and 15 of Treatment
Description: as for outcome 3
Time Frame: Days 7 and 15
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo
Number analyzed (Participants) | 90 | 90
percentage of participants
  Day 7, 1=worse | 2.2 | 0.0
  Day 7, 2=no change | 8.9 | 26.7
  Day 7, 3=slight improvement | 52.2 | 44.4
  Day 7, 4=moderate improvement | 27.8 | 24.4
  Day 7, 5=marked improvement | 8.9 | 4.4
  Day 15, 1=worse | 1.1 | 1.1
  Day 15, 2=no change | 5.6 | 11.1
  Day 15, 3=slight improvement | 27.8 | 34.4
  Day 15, 4=moderate improvement | 30.0 | 32.2
  Day 15, 5=marked improvement | 35.6 | 21.1
Statistical Analysis 1: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; Day 7. The 2-sample Wilcoxon sum rank test was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 0.05 level of significance; Test type: Superiority; p = 0.0330, Wilcoxon Sum Rank Test
Statistical Analysis 2: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; Day 15. The 2-sample Wilcoxon sum rank test was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 0.05 level of significance; Test type: Superiority; p = 0.0262, Wilcoxon Sum Rank Test

5. Secondary Outcome: Percentage of Participants With Subject-Rated Global Impression on Days 3, 7, and 14 of Treatment
Description: Participants assessed their clinical global impression based on relief from local pain, restriction in activities of daily living, restriction of movement and intensity of local pain on a daily basis. The following 5-point rating scale was used: "1 = worse", "2 = no change", "3 = slight improvement", "4 = moderate improvement", "5 = marked improvement".
Time Frame: Days 3, 7, and 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo
Number analyzed (Participants) | 90 | 90
percentage of participants
  Day 3, 1=worse | 3.3 | 1.1
  Day 3, 2=no change | 45.6 | 56.7
  Day 3, 3=slight improvement | 47.8 | 33.3
  Day 3, 4=moderate improvement | 3.3 | 7.8
  Day 3, 5=marked improvement | 0.0 | 1.1
  Day 7, 1=worse | 4.4 | 1.1
  Day 7, 2=no change | 13.3 | 25.6
  Day 7, 3=slight improvement | 52.2 | 43.3
  Day 7, 4=moderate improvement | 22.2 | 25.6
  Day 7, 5=marked improvement | 7.8 | 4.4
  Day 14, 1=worse | 1.1 | 1.1
  Day 14, 2=no change | 14.4 | 26.7
  Day 14, 3=slight improvement | 24.4 | 20.0
  Day 14, 4=moderate improvement | 27.8 | 28.9
  Day 14, 5=marked improvement | 32.2 | 23.3
Statistical Analysis 1: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; Day 3. The 2-sample Wilcoxon sum rank test was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 0.05 level of significance; Test type: Superiority; p = 0.5756, Wilcoxon Sum Rank Test
Statistical Analysis 2: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.4395, Wilcoxon Sum Rank Test
Statistical Analysis 3: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; Day 14. The 2-sample Wilcoxon sum rank test was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 0.05 level of significance; Test type: Superiority; p = 0.0905, Wilcoxon Sum Rank Test

6. Secondary Outcome: Percentage of Responders on Days 3, 7, and 14 of Treatment
Description: A responder was defined as a participant who had both a rating of either "very good" or "excellent" for the participant's rating of medication helpfulness.
Time Frame: Days 3, 7, and 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo
Number analyzed (Participants) | 90 | 90
percentage of participants
  Day 3 | 3.3 | 2.2
  Day 7 | 15.6 | 14.4
  Day 14 | 40.0 | 31.1
Statistical Analysis 1: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; Day 3. A two-tailed Fisher's exact test to compare the number of "responders" between the Placebo and the Cyclobenzaprine HCl 15 mg treatment group to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 0.05 level of significance; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; Day 7. A two-tailed Fisher's exact test to compare the number of "responders" between the Placebo and the Cyclobenzaprine HCl 15 mg treatment group to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 0.05 level of significance; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; Day 14. A two-tailed Fisher's exact test to compare the number of "responders" between the Placebo and the Cyclobenzaprine HCl 15 mg treatment group to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 0.05 level of significance; Test type: Superiority; p = 0.2757, Fisher Exact

7. Secondary Outcome: Percentage of Participants With Physician Rated Assessment of Presence of Muscle Spasm on Days 3, 7, and 15 of Treatment
Description: The investigator assessment based on physical examination, presence of muscle spasm (presence of muscle spasm assessment). The following 5-point rating scale was used: "1 = none", "2 = mild", "3 = moderate", "4 = moderately severe", "5 = severe".
Time Frame: Days 3, 7, and 15
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo
Number analyzed (Participants) | 90 | 90
percentage of participants
  Day 3, 1=none | 2.2 | 2.2
  Day 3, 2=mild | 27.8 | 21.1
  Day 3, 3=moderate | 62.2 | 66.7
  Day 3, 4=moderately severe | 7.8 | 10.0
  Day 3, 5=severe | 0.0 | 0.0
  Day 7, 1=none | 14.4 | 5.6
  Day 7, 2=mild | 47.8 | 53.3
  Day 7, 3=moderate | 37.8 | 38.9
  Day 7, 4=moderately severe | 0.0 | 2.2
  Day 7, 5=severe | 0.0 | 0.0
  Day 15, 1=none | 48.9 | 32.2
  Day 15, 2=mild | 37.8 | 47.8
  Day 15, 3=moderate | 13.3 | 20.0
  Day 15, 4=moderately severe | 0.0 | 0.0
  Day 15, 5=severe | 0.0 | 0.0
Statistical Analysis 1: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.3020, Wilcoxon Sum Rank Test
Statistical Analysis 2: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.2367, Wilcoxon Sum Rank Test
Statistical Analysis 3: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0250, Wilcoxon Sum Rank Test

8. Secondary Outcome: Percentage of Participants With Physician Rated Assessment of Presence of Local Pain on Days 3, 7, and 15 of Treatment
Description: The investigator assessed local pain based on physical examination, reaction to palpation (presence of local pain assessment). The following 5-point rating scale was used: "1 = none", "2 = mild", "3 = moderate", "4 = moderately severe", "5 = severe".
Time Frame: Days 3, 7, and 15
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo
Number analyzed (Participants) | 90 | 90
percentage of participants
  Day 3, 1=none | 1.1 | 1.1
  Day 3, 2=mild | 24.4 | 21.1
  Day 3, 3=moderate | 66.7 | 66.7
  Day 3, 4=moderately severe | 7.8 | 11.1
  Day 3, 5=severe | 0.0 | 0.0
  Day 7, 1=none | 6.7 | 2.2
  Day 7, 2=mild | 55.6 | 50.0
  Day 7, 3=moderate | 36.7 | 46.7
  Day 7, 4=moderately severe | 1.1 | 1.1
  Day 7, 5=severe | 0.0 | 0.0
  Day 15, 1=none | 35.6 | 25.6
  Day 15, 2=mild | 51.1 | 50.0
  Day 15, 3=moderate | 12.2 | 24.4
  Day 15, 4=moderately severe | 1.1 | 0.0
  Day 15, 5=severe | 0.0 | 0.0
Statistical Analysis 1: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.4428, Wilcoxon Sum Rank Test
Statistical Analysis 2: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.1163, Wilcoxon Sum Rank Test
Statistical Analysis 3: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0489, Wilcoxon Sum Rank Test

9. Secondary Outcome: Percentage of Participants With Physician Rated Assessment of Limitation of Range of Motion on Days 3, 7, and 15 of Treatment
Description: The investigator assessed limitation of range of motion. The following 5-point rating scale was used: "1 = none", "2 = mild", "3 = moderate", "4 = moderately severe", "5 = severe".
Time Frame: Days 3, 7, and 15
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo
Number analyzed (Participants) | 90 | 90
percentage of participants
  Day 3, 1=none | 6.7 | 4.4
  Day 3, 2=mild | 40.0 | 37.8
  Day 3, 3=moderate | 47.8 | 52.2
  Day 3, 4=moderately severe | 5.6 | 5.6
  Day 3, 5=severe | 0.0 | 0.0
  Day 7, 1=none | 22.2 | 13.3
  Day 7, 2=mild | 51.1 | 51.1
  Day 7, 3=moderate | 26.7 | 35.6
  Day 7, 4=moderately severe | 0.0 | 0.0
  Day 7, 5=severe | 0.0 | 0.0
  Day 15, 1=none | 44.4 | 38.9
  Day 15, 2=mild | 48.9 | 47.8
  Day 15, 3=moderate | 6.7 | 13.3
  Day 15, 4=moderately severe | 0.0 | 0.0
  Day 15, 5=severe | 0.0 | 0.0
Statistical Analysis 1: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.5275, Wilcoxon Sum Rank Test
Statistical Analysis 2: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0880, Wilcoxon Sum Rank Test
Statistical Analysis 3: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.2542, Wilcoxon Sum Rank Test

10. Secondary Outcome: Percentage of Participants With Physician Rated Assessment of Limitation of Activities of Daily Living on Days 3, 7, and 15 of Treatment
Description: The investigator assessed limitation of activities based on evaluation of the patient's reported functional assessment. The following 5-point rating scale was used: "1 = none", "2 = mild", "3 = moderate", "4 = moderately severe", "5 = severe".
Time Frame: Days 3, 7, and 15
Population: as for outcome 1
Measure: Number; unit: percentage of percentage
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo
Number analyzed (Participants) | 90 | 90
percentage of percentage
  Day 3, 1=none | 4.4 | 5.6
  Day 3, 2=mild | 46.7 | 50.0
  Day 3, 3=moderate | 46.7 | 38.9
  Day 3, 4=moderately severe | 2.2 | 5.6
  Day 3, 5=severe | 0.0 | 0.0
  Day 7, 1=none | 18.9 | 10.0
  Day 7, 2=mild | 62.2 | 63.3
  Day 7, 3=moderate | 17.8 | 26.7
  Day 7, 4=moderately severe | 1.1 | 0.0
  Day 7, 5=severe | 0.0 | 0.0
  Day 15, 1=none | 50.0 | 41.1
  Day 15, 2=mild | 45.6 | 53.3
  Day 15, 3=moderate | 4.4 | 5.6
  Day 15, 4=moderately severe | 0.0 | 0.0
  Day 15, 5=severe | 0.0 | 0.0
Statistical Analysis 1: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.6920, Wilcoxon Sum Rank Test
Statistical Analysis 2: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0749, Wilcoxon Sum Rank Test
Statistical Analysis 3: Comparison: Cyclobenzaprine HCl 15 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.2371, Wilcoxon Sum Rank Test

ADVERSE EVENTS:
Time Frame: First dose of study drug to within 30 days of last dose of study drug (Up to 45 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cyclobenzaprine HCl 15 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 21/90 | 12/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclobenzaprine HCl 15 mg (N=90) | Placebo (N=90)
Tachycardia (Cardiac disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 6 | 1
Flatulence (Gastrointestinal disorders) | 1 | 2
Toothache (Gastrointestinal disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Poor quality sleep (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Disruptive mood dysregulation disorder (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Somnolence (Nervous system disorders) | 18 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT02814565/SAP_000.pdf
  • Study Protocol (2016-08-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT02814565/Prot_001.pdf